CLINICAL TRIAL: NCT02267551
Title: Non-inferiority Study Comparing daVinci Skills Simulator to Mimic dV-Trainer for Preparing Residents to Perform Live Human Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: low enrollment
Sponsor: Atlantic Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Health Services Research
Other Study IDs: 574541-1
Record Dates: First submitted 2014-10-14; First posted 2014-10-17 (Estimated); Last update posted 2016-05-06 (Estimated); Status verified 2016-05

CONDITIONS: Simulation for Preparation of Robotic Surgery
Keywords: robotic surgery; simulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mimic dV-Trainer (Other)
  Interventions: Other: Mimic dv-Trainer
- daVinci Skills Simulator (Other)
  Interventions: Other: daVinci Skills Simulator

INTERVENTIONS:
Other: Mimic dv-Trainer
  Arms: Mimic dV-Trainer
Other: daVinci Skills Simulator
  Arms: daVinci Skills Simulator

SUMMARY:
The objective of this study is to determine whether a group of resident physicians otherwise naïve to robotic surgery can demonstrate equal levels of proficiency during their first robotic supracervical hysterectomy having received training either with the Mimic dV-Trainer or the daVinci Skills Simulator.

ELIGIBILITY:
Inclusion Criteria:

* Obstetrics and gynecology or general surgery residents in ACGME accredited programs naïve to robotic surgery training
* Completion of the online orientation to daVinci Surgical System

Exclusion Criteria:

* Performance of any robotic surgical procedures as the console surgeon
* Performance of any robotic simulator protocols
* Any significant amount of time spent on a virtual reality robotic simulator

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2014-04; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Operative Time | at time of supracervical hysterectomy
  Operative time will be measured by time elapsed between first grasp of the uterine fundus with the robotic single tooth tenaculum until amputation of the specimen at the internal cervical os.

SECONDARY OUTCOMES:
Estimated Blood Loss | during the surgical procedure
  As measured by the blood suctioned into the canister throughout the hysterectomy and at the end of the amputation discounting irrigation volume.
Surgical Skill Rating | following completion of the procedure
  As measured by the global assessment tool for evaluation of intraoperative laparoscopic skills (GOALS) tool via video assessment. These ratings will be performed by a group of surgeons who are not involved in the study and are masked as to the identity of the study surgeons.
Continued success with robotic surgery after participation in the study | during the 12 months following surgical procedure
  The number of cases each participating resident performs as primary surgeon the 12 months after completion of the study will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Morristown Medical Center, Morristown, New Jersey, United States

REFERENCES:
- [Background] Culligan P, Gurshumov E, Lewis C, Priestley J, Komar J, Salamon C. Predictive validity of a training protocol using a robotic surgery simulator. Female Pelvic Med Reconstr Surg. 2014 Jan-Feb;20(1):48-51. doi: 10.1097/SPV.0000000000000045. PMID 24368489